CLINICAL TRIAL: NCT01076023
Title: Comprehensive Cohort Study in Type 2 Diabetes With High Risk of Cardiovascular Disease in China
Brief Title: Cohort Study in Type 2 Diabetes in China
Acronym: CCDC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Cardiometabolic Registries (Network)
Collaborators: Roche Pharma AG (Industry); VitalStrategic Research Institute (Other); Chinese College of Cardiovascular Physicians (Unknown); Chinese Society of Endocrinology (Unknown)
Responsible Party: Sponsor
Other Study IDs: CCMR-301-CCDC; CCDC (Registry Identifier: CCMR)
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Cardiovascular disease; Observational study; China
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is designed to assess the incidence of cardiovascular events occurred within an 12 month follow up period in type 2 diabetic patients with either high risk of cardiovascular disease (CVD) or history of coronary artery disease (CAD) or stroke.

DETAILED DESCRIPTION:
The number of diabetes patients around the world has increased from 30 million in 1985 to the current 180 million, and is expected to grow to 366 million in 2025, with 75 percent occurring in developing countries such as India and China. In China, economic prosperity and changes in diet and lifestyles have resulted in steep increase in prevalence of overweight, obesity, and diabetes. Type 2 diabetes mellitus is associated with an increased risk for both micro-and macrovascular complications, and cardiovascular diseases (CVD) are the most common causes of death in these patients. Preventing the onset or the worsening of the cardiovascular diseases is thus one of the most important goals in managing type II diabetes. This study is designed to better understand the incidence of cardiovascular events under current patterns of treatment in type 2 diabetic patients with either 3 or more risk factors for cardiovascular disease such as older age, hypertension, dyslipidemia, etc, or existing or prior history of coronary artery disease and stroke. Approximately 1000 patients from major hospitals across several regions of China will be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 40 years of age or older
* Patients with confirmed diagnosis of type II diabetes
* Patients with 3 or more CVD risk factors or with confirmed/history of CAD or history of ischemic stroke
* Patients who have lab data within 30 days of baseline visit
* Patients who are willing to return for all follow up visits

Exclusion Criteria:

* Patients who are not willing or not able to return to the same hospital within 12 months after enrollment
* Patients who have life threatening or terminal disease, or are physically unable to make follow up visits every 6 months after enrollment
* Patients have severe heart failure (New York Heart Association [NYHA] Class 3-4)
* Patients with severe renal deficiency (creatinine clearance less than 30 ml/min)
* Patients who are not willing to sign informed consent form

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Out patients of Tier 3 hospitals
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-10 (Actual); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardiovascular events, including fatal and non-fatal acute coronary syndromes (acute myocardial infarction [AMI] or unstable angina), fatal or non-fatal stroke, and other cardiovascular death. | 12 months

SECONDARY OUTCOMES:
Outcomes of current anti-diabetic treatment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, MD, Principal Investigator — Shanghai JiaoTong University RuiJing Hospital
Locations (1):
- Weiqing Wang, Shanghai, Shanghai Municipality, China

REFERENCES:
- See also: Related Info — http://CCMRegistry.org